CLINICAL TRIAL: NCT00191984
Title: Open Multicenter Phase II Study in Second-Line Metastatic Colorectal Cancer Patients: Combination of ALIMTA and Irinotecan Administered Every Two-Weeks
Brief Title: A Study of the Combination of Pemetrexed and Irinotecan Every Two Weeks in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8673; H3E-FP-S057 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-06-15 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Irinotecan (Experimental)
  Interventions: Drug: pemetrexed; Drug: irinotecan

INTERVENTIONS:
Drug: pemetrexed — 400 mg/m^2, intravenous (IV), every 14 days x 12 cycles
  Other Names: LY231514; Alimta
Drug: irinotecan — 180 mg/m^2, intravenous (IV), every 14 days x 12 cycles

SUMMARY:
A non-randomized phase II study to determine the efficacy and safety of the combination of Pemetrexed and Irinotecan every two weeks in metastatic colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal adenocarcinoma that is not amenable to curative therapy.
* Patient must have at least one unidimensionally measurable lesion.
* Prior radiation therapy to less than 25% of bone marrow. Radiation must be completed at least 4 weeks prior to study enrollment.
* Performance status 0 to 2
* Patient must have received 1 prior course of chemotherapy (Folfox regimen) for metastatic disease

Exclusion Criteria:

* Treatment with any drug within the last 30 days that has not received regulatory approval.
* Serious systemic disorder (cardiac or pulmonary disease, active infection)
* Documented brain metastases not amenable to surgery or unstable after radiation
* Inability or unwillingness to take folic acid or Vitamin B12 supplementation.
* Presence of fluid retention that can not be controlled by drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Montfermeil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Suresnes

REFERENCES:
- [Result] Louvet C, Andre T, Gamelin E, Hebbar M, Mabro M, Bennamoun M, Rassam H, de Gramont A. Phase II Study of Biweekly Pemetrexed Plus Irinotecan as Second-Line Therapy for Metastatic Colorectal Cancer. J Oncol. 2010;2010:785934. doi: 10.1155/2010/785934. Epub 2010 Apr 8. PMID 20396391
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants discontinued the trial before receiving study treatment. One due to entry criteria exclusion and one due to withdrawal by subject. Therefore, 44 participants received at least one dose of chemotherapy and are included in the efficacy and safety analyses.
Groups:
- Pemetrexed + Irinotecan: Pemetrexed: 400 mg/m2, intravenous (IV), every 14 days x 12 cycles Irinotecan: 180 mg/m2, intravenous (IV), every 14 days x 12 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Irinotecan
Started | 46
Completed | 7
Not Completed | 39
Not completed — Disease Progression | 21
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Entry Criteria Exclusion | 1
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 31
Region of Enrollment [Number; unit: participants]
  France | 44
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: units on a scale] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  units on a scale
    0 - Fully Active | 24
    1 - Ambulatory, Restricted Strenuous Activity | 15
    2 - Ambulatory, No Work Activities | 5
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma of Colon | 22
  Adenocarcinoma of Rectum | 20
  Colorectal Cancer | 2
Height [Mean (Standard Deviation); unit: centimeters] | 169.3 (8.5)
Weight [Mean (Standard Deviation); unit: kilograms] | 69.3 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
  Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions.
  Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions. Stable disease (SD) = small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 2 years follow-up)
Population: All enrolled participants with at least one completed cycle.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 44
participants
  Partial Response | 6
  Stable Disease | 18
  Progressive Disease | 15
  Unknown | 5

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Response was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
  Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: time of response to progressive disease or death (up to 2 years follow-up)
Population: All enrolled participants with at least completed cycle and who had a complete or partial response.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 6
days | 236 [105 to 353]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from study enrollment to the first date of disease progression or death as a result of any cause. PFS was censored at the date of the last follow-up visit for participants who were still alive and who had not progressed.
Time Frame: baseline to measured progressive disease or death (up to 2 years follow-up)
Population: All enrolled participants with at least one completed cycle.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 44
days | 123 [60 to 146]

4. Secondary Outcome: Time to Treatment Failure
Description: Defined as the time from study enrollment to the first observation of disease progression, death as a result of any cause, or early discontinuation of treatment. Time to treatment failure was censored at the date of the last follow-up visit for patients who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: baseline to stopping treatment (up to 2 years follow-up)
Population: All enrolled participants with at least one completed cycle.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 44
days | 66 [55 to 105]

5. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 2 years follow-up)
Population: All enrolled participants with at least one completed cycle.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Irinotecan
Number analyzed (Participants) | 44
days | 422 [305 to 602]

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Irinotecan
Serious Adverse Events (participants affected / at risk) | 13
Other Adverse Events (participants affected / at risk) | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Irinotecan
Anaemia (Blood and lymphatic system disorders) | 3/44 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1/44 (1)
Diarrhoea (Gastrointestinal disorders) | 3/44 (4)
Melaena (Gastrointestinal disorders) | 1/44 (1)
Nausea (Gastrointestinal disorders) | 1/44 (1)
Vomiting (Gastrointestinal disorders) | 2/44 (2)
Asthenia (General disorders) | 1/44 (1)
General physical health deterioration (General disorders) | 1/44 (1)
Pyrexia (General disorders) | 1/44 (1)
Hepatic pain (Hepatobiliary disorders) | 1/44 (1)
Hypersensitivity (Immune system disorders) | 1/44 (1)
Septic shock (Infections and infestations) | 1/44 (1)
Dehydration (Metabolism and nutrition disorders) | 2/44 (2)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1/44 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1/44 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/44 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/44 (1)
Rash (Skin and subcutaneous tissue disorders) | 1/44 (1)
Hypertensive crisis (Vascular disorders) | 1/44 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Irinotecan
Anaemia (Blood and lymphatic system disorders) | 10/44 (11)
Neutropenia (Blood and lymphatic system disorders) | 7/44 (11)
Conjunctivitis (Eye disorders) | 4/44 (5)
Abdominal pain (Gastrointestinal disorders) | 6/44 (10)
Constipation (Gastrointestinal disorders) | 8/44 (10)
Diarrhoea (Gastrointestinal disorders) | 15/44 (24)
Nausea (Gastrointestinal disorders) | 18/44 (38)
Vomiting (Gastrointestinal disorders) | 11/44 (24)
Asthenia (General disorders) | 24/44 (29)
Mucosal inflammation (General disorders) | 4/44 (10)
Pyrexia (General disorders) | 6/44 (12)
Alanine aminotransferase increased (Investigations) | 4/44 (5)
Aspartate aminotransferase increased (Investigations) | 3/44 (3)
Weight decreased (Investigations) | 9/44 (9)
Weight increased (Investigations) | 3/44 (3)
Anorexia (Metabolism and nutrition disorders) | 8/44 (9)
Anxiety (Psychiatric disorders) | 3/44 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3/44 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days